CLINICAL TRIAL: NCT01663740
Title: A Multicenter Prospective Cohort Study to Investigate if Ganciclovir Significantly Affects Spermatogenesis in Adult Male Renal Transplant Recipients Receiving up to 200 Days Valganciclovir Vs. Concurrent Untreated Matched Controls
Brief Title: A Study on Spermatogenesis in Male Renal Transplant Recipients Receiving Valganciclovir (Valcyte®) Versus Untreated Matched Controls
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Other
Other Study IDs: WV25651
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-07

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

ARMS (2):
- Cohort A: Partcipants who Received Valganciclovir (Experimental): Participants with donor positive (D+)/recipient negative (R-) cytomegalovirus (CMV) serology, who receive valganciclovir prophylaxis according to the local prescribing information, will be observed for spermatogenesis up to 52 weeks post-transplant.
  Interventions: Drug: Valganciclovir
- Cohort B: Untreated Participants (No Intervention): Participants with donor negative (D-)/R- CMV serology, who do not receive prophylaxis, will be observed for spermatogenesis up to 52 weeks post-transplant.

INTERVENTIONS:
Drug: Valganciclovir — Participants will receive valganciclovir 900 milligrams (mg) orally once daily for up to a maximum of 200 days post-transplant.
  Other Names: Valcyte®
  Arms: Cohort A: Partcipants who Received Valganciclovir

SUMMARY:
This observational study will compare spermatogenesis in male adult renal transplant recipients receiving valganciclovir versus untreated matched controls. Data will be collected from each participant for up to 52 weeks post transplant.

ELIGIBILITY:
Inclusion Criteria:

* First renal transplant
* Participant eligible to receive valganciclovir prophylaxis as determined by the treating physician in accordance with the local approved product prescribing information (Cohort A only) or the participant is not expected to require any valganciclovir prophylaxis (Cohort B only) post-transplant
* Participant has no history of known infertility
* Participant is able and willing to provide semen samples
* Participant agrees to utilize a barrier contraceptive throughout the study or for at least 90 days after cessation of valganciclovir treatment

Exclusion Criteria:

* Prior ganciclovir or valganciclovir within 3 months of enrollment
* Organ transplant other than kidney
* Participant has received an investigational new drug in the 3 months prior to transplant
* Participant hs received an alkylating agent or other medications known to affect fertility/spermatogenesis
* Participant is unlikely to be available for follow-up for the entire duration of the study (up to 52 weeks)

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2012-01-30 (Actual); Primary Completion 2015-09-29 (Actual); Study Completion 2016-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- United States (16):
  - National Institute of Transplantation, Los Angeles, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Medical College of Georgia, Augusta, Georgia
  - Tufts Medical Center, Boston, Massachusetts
  - Western New England Renal & Transplant Associates, P.C., Springfield, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Albany Medical Cancer Center, Albany, New York
  - University at Buffalo, Buffalo, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Oregan Health & Science Univ, Portland, Oregon
  - Drexel University Department of Nephrology, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
- Mexico (3):
  - Hospital Miguel Hidalgo, Aguascalientes
  - Instituto Mexicano de Trasplantes, Cuernavaca
  - Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Partcipants Who Received Valganciclovir: Participants with donor positive (D+)/recipient negative (R-) cytomegalovirus (CMV) serology, who received valganciclovir prophylaxis according to the local prescribing information, were observed for spermatogenesis up to 52 weeks post-transplant.
- Cohort B: Untreated Participants: Participants with donor negative (D-)/R- CMV serology, who did not receive prophylaxis, were observed for spermatogenesis up to 52 weeks post-transplant.
Period: Overall Study
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Started | 38 (Safety Population) | 21 (Safety Population)
Completed | 22 | 13
Not Completed | 16 | 8
Not completed — Lost to Follow-up | 1 | 4
Not completed — Other | 9 | 2
Not completed — Inclusion/Exclusion not met | 1 | 0
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — No end of study status | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants assigned to a cohort. One participant who was considered for inclusion in the study but did not participate, was excluded from baseline analysis.
Groups:
- Cohort A: Partcipants Who Received Valganciclovir: Participants with D+/R- CMV serology, who received valganciclovir prophylaxis according to the local prescribing information, were observed for spermatogenesis up to 52 weeks post-transplant.
- Cohort B: Untreated Participants: Participants with D-/R- CMV serology, who did not receive prophylaxis, were observed for spermatogenesis up to 52 weeks post-transplant.
- Total: Total of all reporting groups
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants | Total
Number analyzed (Participants) | 37 | 21 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (7.96) | 32.5 (5.81) | 34.5 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 37 | 21 | 58
Seminal Volume [Mean (Standard Deviation); unit: milliliters (mL)] — Population: Number analyzed indicates number of participants evaluated for this analysis.
  milliliters (mL)
    number analyzed (Participants) | 30 | 20 | 50
    (all) | 2.4 (1.51) | 2.0 (1.37) | 2.2 (1.46)
Sperm Density [Mean (Standard Deviation); unit: millions of sperm/milliliter (mil/mL)] — Population: Number analyzed indicates number of participants evaluated for this analysis.
  millions of sperm/milliliter (mil/mL)
    number analyzed (Participants) | 30 | 20 | 50
    (all) | 21.0 (28.33) | 23.2 (24.90) | 21.9 (26.77)
Percentage of Normal Sperm Cells [Mean (Standard Deviation); unit: percentage of normal sperm cells] — Population: Number analyzed indicates number of participants evaluated for this analysis.
  percentage of normal sperm cells
    number analyzed (Participants) | 27 | 18 | 45
    (all) | 11.4 (18.44) | 33.5 (39.03) | 20.3 (30.15)
Total Motility of Sperm [Mean (Standard Deviation); unit: percent motility] — Population: Number analyzed indicates number of participants evaluated for this analysis.
  percent motility
    number analyzed (Participants) | 30 | 20 | 50
    (all) | 25.8 (20.46) | 36.3 (24.24) | 30.0 (22.42)
Terminal Uridine Nick-End Labeling (TUNEL) Score [Mean (Standard Deviation); unit: units on a scale] — TUNEL score represents percentage of sperm with fragmented Deoxyribonucleic acid (DNA); total score ranged from 0 percent (%) to 100%, higher score represents more fragmentation. Population: Number analyzed indicates number of participants evaluated for this analysis.
  units on a scale
    number analyzed (Participants) | 28 | 18 | 46
    (all) | 14.4 (9.80) | 12.9 (10.60) | 13.8 (10.03)
Follicle Stimulating Hormone (FSH) Level [Mean (Standard Deviation); unit: units per liter (U/L)] — Population: Number analyzed indicates number of participants evaluated for this analysis.
  units per liter (U/L)
    number analyzed (Participants) | 29 | 20 | 49
    (all) | 10.8 (6.77) | 8.6 (6.61) | 9.9 (6.72)
Luteinizing Hormone (LH) Level [Mean (Standard Deviation); unit: milliunits per milliliter (mU/mL)] — Population: Number analyzed indicates number of participants evaluated for this analysis.
  milliunits per milliliter (mU/mL)
    number analyzed (Participants) | 29 | 20 | 49
    (all) | 6.4 (2.61) | 6.8 (6.86) | 6.6 (4.76)
Prolactin Level [Mean (Standard Deviation); unit: mU/mL] — Population: Number analyzed indicates number of participants evaluated for this analysis.
  mU/mL
    number analyzed (Participants) | 29 | 20 | 49
    (all) | 175.4 (73.51) | 164.5 (46.22) | 170.9 (63.46)
Testosterone Level [Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)] — Population: Number analyzed indicates number of participants evaluated for this analysis.
  nanomoles per liter (nmol/L)
    number analyzed (Participants) | 29 | 20 | 49
    (all) | 14.2 (5.83) | 11.3 (5.54) | 13.0 (5.84)
Inhibin B Level [Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)] — Population: Number analyzed indicates number of participants evaluated for this analysis.
  picograms per milliliter (pg/mL)
    number analyzed (Participants) | 27 | 19 | 46
    (all) | 103.4 (55.82) | 149.1 (98.45) | 122.3 (78.70)

OUTCOME MEASURES:

1. Primary Outcome: Change in Sperm Density From Baseline to the End of Treatment (EOT)
Description: Sperm density was calculated based on the average of two semen samples. Change was calculated as the sperm density measured at post-baseline visit (EOT) minus (-) the sperm density measured at baseline for each participant. A negative change from baseline indicated a lower sperm density (worsening).
Time Frame: Baseline, EOT (Week 28)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: mil/mL
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 24 | 14
mil/mL | -9.770 (9.0518) | 30.396 (11.3044)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.0075, Mixed Models Analysis; Model adjusted for Cohort,visit,Cohort by visit interaction,baseline sperm density,age,& duration of pre-transplant dialysis as explanatory variables; Mean Difference = -40.166, 95% CI 2-sided [-68.869 to -11.463], Standard Error of Mean 14.1387 — Change in sperm density from Baseline to EOT

2. Secondary Outcome: Change in Terminal Uridine Nick-End Labeling (TUNEL) Score From Baseline to EOT and End of Follow-up (FU)
Description: Sperm DNA fragmentation change (chromatin damage) was evaluated based on TUNEL score. Change was calculated as the TUNEL score measured at post-baseline visit (EOT and FU) minus the TUNEL score measured at baseline for each participant. A negative change from baseline indicated a lower TUNEL score. TUNEL score represents percentage of sperm with fragmented DNA; total score ranged from 0 percent (%) to 100%, higher score represents more fragmentation.
Time Frame: Baseline, EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure. Number analyzed indicates number of participants evaluated for this outcome measure at specified timepoint.
Measure: Mean (Standard Error); unit: percent score
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 22 | 14
percent score
  Change at EOT | -3.595 (1.7720) | -5.354 (2.0680)
  Change at end of FU: number analyzed (Participants) | 18 | 10
  Change at end of FU | -4.516 (1.9542) | -3.465 (2.5475)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.5109, Mixed Models Analysis; Model adjusted for Cohort,visit,Cohort by visit interaction,baseline TUNEL score,age,& duration of pre-transplant dialysis as explanatory variables; Mean Difference = 1.758, 95% CI 2-sided [-3.619 to 7.135], Standard Error of Mean 2.6460 — Change in TUNEL score from Baseline to EOT
Statistical Analysis 2: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.7449, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference = -1.051, 95% CI 2-sided [-7.566 to 5.464], Standard Error of Mean 3.2058 — Change in TUNEL score from Baseline to end of FU

3. Secondary Outcome: Change in TUNEL Score From EOT to End of FU
Description: Sperm DNA fragmentation change (chromatin damage) was evaluated based on TUNEL score. Change was calculated as the TUNEL score measured at FU minus the TUNEL score measured at EOT for each participant. A negative change from EOT indicated a lower TUNEL score. TUNEL score represents percentage of sperm with fragmented DNA; total score ranged from 0% to 100%, higher score represents more fragmentation.
Time Frame: EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: percent score
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 16 | 9
percent score | 4.447 (2.0671) | 1.578 (2.5315)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.3940, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference = 2.869, 95% CI 2-sided [-4.001 to 9.739], Standard Error of Mean 3.2934 — Change in TUNEL score from EOT to end of FU

4. Secondary Outcome: Change in Seminal Volume From Baseline to EOT and End of FU
Description: Seminal volume was calculated based on the average of two semen samples. Change was calculated as the seminal volume measured at post-baseline visit (EOT and FU) - the seminal volume measured at baseline for each participant. A negative change from baseline indicated a lower seminal volume (worsening).
Time Frame: Baseline, EOT (Week 28), end of FU (Week 52)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mL
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 25 | 14
mL
  Change at EOT | -0.193 (0.2324) | -0.347 (0.2967)
  Change at end of FU: number analyzed (Participants) | 20 | 10
  Change at end of FU | -0.289 (0.2066) | -0.161 (0.2685)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.6773, Mixed Models Analysis; Model adjusted for Cohort,visit,Cohort by visit interaction,baseline semen volume,age,& duration of pre-transplant dialysis as explanatory variables; Mean Difference = 0.155, 95% CI 2-sided [-0.594 to 0.903], Standard Error of Mean 0.3687 — Change in seminal volume from Basline to EOT
Statistical Analysis 2: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.7046, Mixed Models Analysis; [statistical method as in outcome 4, analysis 1]; Mean Difference = -0.128, 95% CI 2-sided [-0.806 to 0.551], Standard Error of Mean 0.3343 — Change in seminal volume from Baseline to end of FU

5. Secondary Outcome: Change in Seminal Volume From EOT to End FU
Description: Seminal volume was calculated based on the average of two semen samples. Change was calculated as the seminal volume measured at FU - the seminal volume measured at EOT for each participant. A negative change from EOT indicated a lower seminal volume (worsening).
Time Frame: EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: mL
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 20 | 9
mL | -0.103 (0.2187) | 0.024 (0.3067)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.7323, Mixed Models Analysis; [statistical method as in outcome 4, analysis 1]; Mean Difference = -0.128, 95% CI 2-sided [-0.888 to 0.633], Standard Error of Mean 0.3684 — Change in seminal volume from EOT to end of FU

6. Secondary Outcome: Change in Sperm Density From EOT to End of FU
Description: Sperm density was calculated based on the average of two semen samples. Change was calculated as the sperm density measured at FU - the sperm density measured at EOT for each participant. A negative change from EOT indicated a lower sperm density (worsening).
Time Frame: EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: mil/mL
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 19 | 9
mil/mL | 57.149 (17.7736) | 5.882 (27.4837)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.1756, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference = 51.267, 95% CI 2-sided [-24.626 to 127.159], Standard Error of Mean 36.6869 — Change in sperm density from EOT to end of FU

7. Secondary Outcome: Change in Sperm Density From Baseline to End of FU
Description: Sperm density was calculated based on the average of two semen samples. Change was calculated as the sperm density measured at post-baseline visit (FU) - the sperm density measured at baseline for each participant. A negative change from baseline indicated a lower sperm density (worsening).
Time Frame: Baseline, end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: mil/mL
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 20 | 10
mil/mL | 39.671 (11.6679) | 49.866 (15.8282)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.6058, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference = -10.195, 95% CI 2-sided [-49.934 to 29.543], Standard Error of Mean 19.5745 — Change in sperm density from Baseline to end of FU

8. Secondary Outcome: Change in Total Motility of Sperm From Baseline to EOT and End of FU
Description: Sperm motility was calculated based on the average of two semen samples. Percent was determined by the calculation of motile sperm/total sperm count. Change was calculated as the sperm motility measured at post-baseline visit (EOT and FU) - the sperm motility measured at baseline for each participant. A negative change from baseline indicated a lower sperm motility (worsening).
Time Frame: Baseline, EOT (Week 28), end of FU (Week 52)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percent motility
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 24 | 14
percent motility
  Change at EOT | 3.839 (5.4259) | 25.667 (6.9723)
  Change at FU: number analyzed (Participants) | 20 | 10
  Change at FU | 24.736 (4.7920) | 34.538 (6.6024)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.0222, Mixed Models Analysis; Model adjusted for Cohort,visit,Cohort by visit interaction,baseline sperm motility,age,duration of pre-transplant dialysis as explanatory variables; Mean Difference = -21.828, 95% CI 2-sided [-40.346 to -3.311], Standard Error of Mean 9.1214 — Change in total motility of sperm from Baseline to EOT
Statistical Analysis 2: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.2495, Mixed Models Analysis; [statistical method as in outcome 8, analysis 1]; Mean Difference = -9.802, 95% CI 2-sided [-26.795 to 7.190], Standard Error of Mean 8.3702 — Change in total motility of sperm from Baseline to end of FU

9. Secondary Outcome: Change in Total Motility of Sperm From EOT to End of FU
Description: Sperm motility was calculated based on the average of two semen samples. Percent was determined by the calculation of motile sperm/total sperm count. Change was calculated as the sperm motility measured at FU - the sperm motility measured at EOT for each participant. A negative change from EOT indicated a lower sperm motility (worsening).
Time Frame: EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: percent motility
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 19 | 9
percent motility | 8.953 (6.3968) | 20.635 (9.0663)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.3505, Mixed Models Analysis; [statistical method as in outcome 8, analysis 1]; Mean Difference = -11.683, 95% CI 2-sided [-37.039 to 13.674], Standard Error of Mean 12.2576 — Change in total motility of sperm from EOT to end of FU

10. Secondary Outcome: Change in Sperm Morphology Evaluated as Percentage of Normal Sperm Cells From Baseline to EOT and End of FU
Description: Sperm morphology was evaluated based on the average of two semen samples. Change was calculated as the sperm morphology measured at post-baseline visit (EOT and FU) - the sperm morphology measured at baseline for each participant. A positive change from baseline indicated an improved sperm morphology.
Time Frame: Baseline, EOT (Week 28), end of FU (Week 52)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage of normal sperm cells
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 21 | 12
percentage of normal sperm cells
  Change at EOT | 3.720 (4.0233) | 9.461 (5.2737)
  Change at end of FU: number analyzed (Participants) | 19 | 8
  Change at end of FU | 5.128 (2.8907) | 6.982 (4.2060)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.4021, Mixed Models Analysis; Model adjusted for Cohort,visit,Cohort by visit interaction,baseline sperm morphology,age,pre-transplant dialysis duration as explanatory variables; Mean Difference = -5.741, 95% CI 2-sided [-19.524 to 8.042], Standard Error of Mean 6.7578 — Change in sperm morphology from Baseline to EOT
Statistical Analysis 2: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.7229, Mixed Models Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference = -1.854, 95% CI 2-sided [-12.423 to 8.714], Standard Error of Mean 5.1817 — Change in sperm morphology from Baseline to end of FU

11. Secondary Outcome: Change in Sperm Morphology Evaluated as Percentage of Normal Sperm Cells From EOT to End of FU
Description: Sperm morphology was evaluated based on the average of two semen samples. Change was calculated as the sperm morphology measured at FU - the sperm morphology measured at EOT for each participant. A positive change from EOT indicated an improved sperm morphology.
Time Frame: EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: percentage of normal sperm cells
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 17 | 7
percentage of normal sperm cells | -0.714 (4.3420) | 2.236 (5.8507)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.7080, Mixed Models Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference = -2.950, 95% CI 2-sided [-19.192 to 13.291], Standard Error of Mean 7.7598 — Change in sperm morphology from EOT to end of FU

12. Secondary Outcome: Change in Total Testosterone Level From Baseline to EOT and End of FU
Description: Testosterone level was calculated based on the average of two samples. Change was calculated as the testosterone level measured at post-baseline visit (EOT and FU) - the testosterone level measured at baseline for each participant. A negative change from baseline indicated a lower testosterone level.
Time Frame: Baseline, EOT (Week 28), end of FU (Week 52)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 26 | 14
nmol/L
  Change at EOT | 0.762 (1.0203) | 2.623 (1.3586)
  Change at end of FU: number analyzed (Participants) | 19 | 11
  Change at end of FU | 0.395 (1.0260) | 1.509 (1.3074)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.2673, Mixed Models Analysis; Model adjusted for Cohort,visit,Cohort by visit interaction,baseline testosterone,age,duration of pre-transplant dialysis as explanatory variables; Mean Difference = -1.861, 95% CI 2-sided [-5.213 to 1.491], Standard Error of Mean 1.6512 — Change in total testosterone level from Baseline to EOT
Statistical Analysis 2: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.4949, Mixed Models Analysis; [statistical method as in outcome 12, analysis 1]; Mean Difference = -1.114, 95% CI 2-sided [-4.392 to 2.164], Standard Error of Mean 1.6147 — Change in total testosterone level from Baseline to end of FU

13. Secondary Outcome: Change in Total Testosterone Level From EOT to End of FU
Description: Testosterone level was calculated based on the average of two samples. Change was calculated as the testosterone level measured at FU - the testosterone level measured at EOT for each participant. A negative change from EOT indicated a lower testosterone level.
Time Frame: EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 19 | 11
nmol/L | -0.936 (0.9950) | -0.984 (1.2012)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.9753, Mixed Models Analysis; [statistical method as in outcome 12, analysis 1]; Mean Difference = 0.047, 95% CI 2-sided [-3.063 to 3.157], Standard Error of Mean 1.5100 — Change in total testosterone level from EOT to end of FU

14. Secondary Outcome: Change in LH Level From Baseline to EOT and End of FU
Description: LH level was calculated based on the average of two samples. Change was calculated as the LH level measured at post-baseline visit (EOT and FU) - the LH level measured at baseline for each participant. A negative change from baseline indicated a lower LH level.
Time Frame: Baseline, EOT (Week 28), end of FU (Week 52)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mU/mL
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 26 | 13
mU/mL
  Change at EOT | -0.281 (0.3743) | -0.357 (0.5190)
  Change at end of FU: number analyzed (Participants) | 20 | 11
  Change at end of FU | -1.857 (0.2787) | -0.642 (0.3635)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.9053, Mixed Models Analysis; Model adjusted for Cohort,visit,Cohort by visit interaction,baseline LH concentration,age,pre-transplant dialysis duration as explanatory variables; Mean Difference = 0.076, 95% CI 2-sided [-1.214 to 1.366], Standard Error of Mean 0.6347 — Change in LH level from Baseline to EOT
Statistical Analysis 2: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.0104, Mixed Models Analysis; [statistical method as in outcome 14, analysis 1]; Mean Difference = -1.215, 95% CI 2-sided [-2.125 to -0.305], Standard Error of Mean 0.4477 — Change in LH level from Baseline to end of FU

15. Secondary Outcome: Change in LH Level From EOT to End of FU
Description: LH level was calculated based on the average of two samples. Change was calculated as the LH level measured at FU - the LH level measured at EOT for each participant. A negative change from EOT indicated a lower LH level.
Time Frame: EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: mU/mL
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 20 | 11
mU/mL | -1.482 (0.2607) | -0.417 (0.3207)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.0143, Mixed Models Analysis; Model adjusted for Cohort,visit,Cohort by visit interaction,baseline LH concentration,age,& pre-transplant dialysis duration as explanatory variables; Mean Difference = -1.065, 95% CI 2-sided [-1.899 to -0.231], Standard Error of Mean 0.4057 — Change in LH level from EOT to end of FU

16. Secondary Outcome: Change in FSH Level From Baseline to EOT and End of FU
Description: FSH level was calculated based on the average of two samples. Change was calculated as the FSH level measured at post-baseline visit (EOT and FU) - the FSH level measured at baseline for each participant. A negative change from baseline indicated a lower FSH level.
Time Frame: Baseline, EOT (Week 28), end of FU (Week 52)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 26 | 13
U/L
  Change at EOT | 1.521 (1.0033) | -1.020 (1.4072)
  Change at end of FU: number analyzed (Participants) | 20 | 11
  Change at end of FU | -2.905 (0.4113) | -1.922 (0.5369)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.1505, Mixed Models Analysis; Model adjusted for Cohort,visit,Cohort by visit interaction,baseline FSH concentration,age,pre-transplant dialysis duration as explanatory variables; Mean Difference = 2.541, 95% CI 2-sided [-0.969 to 6.052], Standard Error of Mean 1.7274 — Change in FSH level from Baseline to EOT
Statistical Analysis 2: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.1539, Mixed Models Analysis; [statistical method as in outcome 16, analysis 1]; Mean Difference = -0.983, 95% CI 2-sided [-2.352 to 0.387], Standard Error of Mean 0.6739 — Change in FSH level from Baseline to end of FU

17. Secondary Outcome: Change in FSH Level From EOT to End of FU
Description: FSH level was calculated based on the average of two samples. Change was calculated as the FSH level measured at FU - the FSH level measured at EOT for each participant. A negative change from EOT indicated a lower FSH level.
Time Frame: EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 20 | 11
U/L | -3.462 (0.5036) | -1.988 (0.6141)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.0798, Mixed Models Analysis; [statistical method as in outcome 16, analysis 1]; Mean Difference = -1.474, 95% CI 2-sided [-3.136 to 0.188], Standard Error of Mean 0.8084 — Change in FSH level from EOT to end of FU

18. Secondary Outcome: Change in Prolactin Level From Baseline to EOT and End of FU
Description: Prolactin level was calculated based on the average of two samples. Change was calculated as the prolactin level measured at post-baseline visit (EOT and FU) - the prolactin level measured at baseline for each participant. A negative change from baseline indicated a lower prolactin level.
Time Frame: Baseline, EOT (Week 28), end of FU (Week 52)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mU/mL
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 25 | 13
mU/mL
  Change at EOT | 15.590 (14.4761) | 15.693 (19.2663)
  Change at end of FU: number analyzed (Participants) | 20 | 11
  Change at end of FU | 9.829 (13.1691) | -5.443 (16.7203)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.9965, Mixed Models Analysis; Model adjusted for Cohort,visit,Cohort by visit interaction,baseline prolactin level,age,pre-transplant dialysis duration as explanatory variables; Mean Difference = -0.104, 95% CI 2-sided [-47.792 to 47.585], Standard Error of Mean 23.4660 — Change in prolactin level from Baseline to EOT
Statistical Analysis 2: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.4636, Mixed Models Analysis; [statistical method as in outcome 18, analysis 1]; Mean Difference = 15.272, 95% CI 2-sided [-26.599 to 57.142], Standard Error of Mean 20.6031 — Change in prolactin level from Baseline to end of FU

19. Secondary Outcome: Change in Prolactin Level From EOT to End of FU
Description: Prolactin level was calculated based on the average of two samples. Change was calculated as the prolactin level measured at FU - the prolactin level measured at EOT for each participant. A negative change from EOT indicated a lower prolactin level.
Time Frame: EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: mU/mL
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 19 | 11
mU/mL | -7.429 (10.9988) | -16.169 (13.5322)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.6134, Mixed Models Analysis; [statistical method as in outcome 18, analysis 1]; Mean Difference = 8.740, 95% CI 2-sided [-26.438 to 43.917], Standard Error of Mean 17.0805 — Change in prolactin level from EOT to end of FU

20. Secondary Outcome: Change in Inhibin B Level From Baseline to EOT and End of FU
Description: Inhibin B level was calculated based on the average of two samples. Change was calculated as the inhibin B level measured at post-baseline visit (EOT and FU) - the inhibin B level measured at baseline for each participant. A negative change from baseline indicated a lower inhibin B level.
Time Frame: Baseline, EOT (Week 28), end of FU (Week 52)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 22 | 12
pg/mL
  Change at EOT | 5.075 (7.3778) | -3.067 (9.5924)
  Change at end of FU: number analyzed (Participants) | 17 | 10
  Change at end of FU | 51.416 (10.8658) | 10.734 (13.9963)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.5002, Mixed Models Analysis; Model adjusted for Cohort,visit,Cohort by visit interaction,baseline inhibin B level,age,pre-transplant dialysis duration as explanatory variables; Mean Difference = 8.142, 95% CI 2-sided [-16.223 to 32.506], Standard Error of Mean 11.9301 — Change in inhibin B level from Baseline to EOT
Statistical Analysis 2: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.0279, Mixed Models Analysis; [statistical method as in outcome 20, analysis 1]; Mean Difference = 40.682, 95% CI 2-sided [4.720 to 76.643], Standard Error of Mean 17.6084 — Change in inhibin B level from Baseline to end of FU

21. Secondary Outcome: Change in Inhibin B Level From EOT to End of FU
Description: Inhibin B level was calculated based on the average of two samples. Change was calculated as the inhibin B level measured at FU - the inhibin B level measured at EOT for each participant. A negative change from EOT indicated a lower inhibin B level.
Time Frame: EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 18 | 9
pg/mL | 40.329 (13.8221) | 14.448 (17.8932)
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; p = 0.2548, Mixed Models Analysis; [statistical method as in outcome 20, analysis 1]; Mean Difference = 25.881, 95% CI 2-sided [-20.024 to 71.786], Standard Error of Mean 22.1348 — Change in inhibin B level from EOT to end of FU

22. Secondary Outcome: Percentage of Participants With Abnormal Sperm Density (<20 Mil/mL) From Baseline to EOT and End of FU
Description: Abnormal sperm density was considered as sperm density less than (<) 20 mil/mL. Change in abnormal to abnormal sperm density and normal to abnormal sperm density from baseline to EOT and end of FU was reported.
Time Frame: Baseline, EOT (Week 28), end of FU (Week 52)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 24 | 14
percentage of participants
  Abnormal to abnormal: EOT | 50.0 | 35.7
  Abnormal to abnormal: FU: number analyzed (Participants) | 20 | 10
  Abnormal to abnormal: FU | 25.0 | 20.0
  Normal to abnormal: EOT | 25.0 | 7.1
  Normal to abnormal: FU: number analyzed (Participants) | 20 | 10
  Normal to abnormal: FU | 0.0 | 0.0
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; Difference in Percentage = 14.3, 95% CI 2-sided [-19.3 to 45.3] — Change in abnormal to abnormal sperm density from Baseline to EOT
Statistical Analysis 2: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; Difference in Percentage = 5.0, 95% CI 2-sided [-34.3 to 43.3] — Change in abnormal to abnormal sperm density from Baseline to end of FU
Statistical Analysis 3: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; Difference in Percentage = 17.9, 95% CI 2-sided [-15.3 to 48.8] — Change in normal to abnormal sperm density from Baseline to EOT

23. Secondary Outcome: Percentage of Participants With Abnormal Sperm Density (<20 Mil/mL) From EOT to End of FU
Description: Abnormal sperm density was considered as sperm density <20 mil/mL. Change in abnormal to abnormal sperm density and normal to abnormal sperm density from EOT to end of FU was reported.
Time Frame: EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 19 | 9
percentage of participants
  Abnormal to abnormal | 26.3 | 22.2
  Normal to abnormal | 0.0 | 0.0
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; Difference in Percentage = 4.1, 95% CI 2-sided [-34.5 to 42.5] — Change in abnormal to abnormal sperm density from EOT to end of FU

24. Secondary Outcome: Percentage of Participants With Improved TUNEL Score From Baseline to EOT and End of FU
Description: Sperm DNA fragmentation change (chromatin damage) was evaluated based on TUNEL score. Participants who had a lower TUNEL score compared to the previous time point were considered as improved.
Time Frame: Baseline, EOT (Week 28), end of FU (Week 52)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 22 | 14
percentage of participants
  EOT | 72.7 | 71.4
  FU: number analyzed (Participants) | 18 | 10
  FU | 66.7 | 60.0
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; Difference in Percentage = 1.3, 95% CI 2-sided [-31.3 to 33.7] — Improvement from Baseline to EOT
Statistical Analysis 2: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; Difference in Percentage = 6.7, 95% CI 2-sided [-31.1 to 44.4] — Improvement from Baseline to end of FU

25. Secondary Outcome: Percentage of Participants With Improved TUNEL Score From EOT to End of FU
Description: as for outcome 24
Time Frame: EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 16 | 9
percentage of participants | 43.8 | 55.6
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; Difference in Percentage = -11.8, 95% CI 2-sided [-50.0 to 29.3] — Improvement from EOT to end of FU

26. Secondary Outcome: Percentage of Participants With Improved Sperm Density From Baseline to EOT and End of FU
Description: Participants who had higher sperm density compared with the previous visit were considered as improved.
Time Frame: Baseline, EOT (Week 28), end of FU (Week 52)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 24 | 14
percentage of participants
  EOT | 33.3 | 64.3
  FU: number analyzed (Participants) | 20 | 10
  FU | 90.0 | 80.0
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; Difference in Percentage = -31.0, 95% CI 2-sided [-59.7 to 2.7] — Improvement from Baseline to EOT
Statistical Analysis 2: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; Difference in Percentage = 10.0, 95% CI 2-sided [-29.7 to 47.7] — Improvement from Baseline to end of FU

27. Secondary Outcome: Percentage of Participants With Improved Sperm Density From EOT to End of FU
Description: Participants who had higher sperm density compared with the previous visit were considered as improved.
Time Frame: EOT (Week 28), end of FU (Week 52)
Population: Safety population. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Number analyzed (Participants) | 19 | 9
percentage of participants | 78.9 | 88.9
Statistical Analysis 1: Comparison: Cohort A: Partcipants Who Received Valganciclovir vs Cohort B: Untreated Participants; Test type: Superiority or Other; Difference in Percentage = -9.9, 95% CI 2-sided [-47.2 to 27.9] — Improvement from EOT to end of FU

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (Week 52)
Description: Participants who received at least one dose of valganciclovir in Cohort A and all transplanted participants of Cohort B were included for adverse events analysis.
Arm/Group | Cohort A: Partcipants Who Received Valganciclovir | Cohort B: Untreated Participants
Serious Adverse Events (participants affected / at risk) | 10/31 | 12/21
Other Adverse Events (participants affected / at risk) | 24/31 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Partcipants Who Received Valganciclovir (N=31) | Cohort B: Untreated Participants (N=21)
Transplant rejection (Immune system disorders) | 3 | 1
Kidney transplant rejection (Immune system disorders) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Retroperitoneal hematoma (Gastrointestinal disorders) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 3
Death (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Perinephric collection (Injury, poisoning and procedural complications) | 0 | 1
Fetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Treatment noncompliance (Social circumstances) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Partcipants Who Received Valganciclovir (N=31) | Cohort B: Untreated Participants (N=21)
Anaemia (Blood and lymphatic system disorders) | 7 | 5
Leukopenia (Blood and lymphatic system disorders) | 6 | 4
Polycythaemia (Blood and lymphatic system disorders) | 2 | 1
Incision site pain (Injury, poisoning and procedural complications) | 4 | 12
Procedural pain (Injury, poisoning and procedural complications) | 2 | 2
Incision site haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Perinephric collection (Injury, poisoning and procedural complications) | 2 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2
Tremor (Nervous system disorders) | 7 | 5
Headache (Nervous system disorders) | 3 | 4
Hypoaesthesia (Nervous system disorders) | 2 | 1
Paraesthesia (Nervous system disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 2
Blood creatinine increased (Investigations) | 6 | 4
Transaminases increased (Investigations) | 5 | 2
Immunosuppressant drug level increased (Investigations) | 0 | 4
Blood pressure increased (Investigations) | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 3 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 4 | 5
Dysuria (Renal and urinary disorders) | 1 | 4
Hydronephrosis (Renal and urinary disorders) | 3 | 0
Proteinuria (Renal and urinary disorders) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 1 | 3
Escherichia infection (Infections and infestations) | 0 | 3
Staphylococcal infection (Infections and infestations) | 2 | 0
Pyrexia (General disorders) | 3 | 4
Oedema peripheral (General disorders) | 5 | 0
Fatigue (General disorders) | 4 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypertension (Vascular disorders) | 3 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 2
Transplant rejection (Immune system disorders) | 3 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Scrotal swelling (Reproductive system and breast disorders) | 2 | 0
Wound drainage (Surgical and medical procedures) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.